CLINICAL TRIAL: NCT00468403
Title: Islet Transplantation in Type I Diabetes With LEA29Y (Belatacept) Maintenance Therapy (CIT-04)
Brief Title: LEA29Y (Belatacept) Emory Edmonton Protocol
Acronym: LEEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Islet Transplantation Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-04
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin dependence; Hypoglycemia; Hypoglycemia unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Abatacept; Basiliximab; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Pancreatic Islet Cells (Experimental): Participants will receive up to three islet transplantations and continuous immunosuppressive therapy including belatacept
  Interventions: Biological: Allogeneic Pancreatic Islet Cells; Biological: Belatacept; Biological: Basiliximab; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Procedure: Intraportal infusion of islet cells

INTERVENTIONS:
Biological: Allogeneic Pancreatic Islet Cells — Transplant of islet cells from a healthy pancreas. A dose of at least 5,000 Islet Equivalents (IEQ)/kg recipient body weight (BW) infused intraportally for the first transplant, and at least 4,000 IEQ/kg recipient BW infused intraportally for subsequent transplants.
Biological: Belatacept — Belatacept is an inhibitor of the 2 signals that stimulate T-cells. Subjects will receive NULOJIX® (belatacept)10mg/kg through a peripheral vein on Day 0 and post-operative days 4, 14, 28, 56, 84. After Day 84 subjects will receive belatacept at a maintenance dose of 5 mg/kg every 4 weeks for the duration of study follow-up (2 years after the final islet transplant). Infusion doses will be based upon the subject's actual body weight at study Day 0 and will not be modified during the course of the study unless there is a change in body weight plus or minus 10% of Day 0 body weight.
  Other Names: NUJOLIX
Biological: Basiliximab — Immunosuppressive medication for prophylaxis of acute transplant rejection. Two Intravenous (IV) doses of basiliximab, a monoclonal antibody Interleukin 2 (IL-2) receptor blocker, will be given with the first and second (if necessary) transplants. The first dose will be 20 mg and will be given within two hours prior to islet transplant on the day of islet transplantation. The second 20 mg dose will be given on Day 4 after the transplant.If a third islet transplant is deemed necessary and performed more than 70 days after the second transplant, both doses of basiliximab will be repeated. No additional doses of basiliximab will be given with a third transplant that is performed between 30 and 70 days after the second transplant.
  Other Names: Simulect
Drug: Mycophenolate Mofetil — Maintenance immunosuppressive therapy. Subjects will receive mycophenolate mofetil starting immediately pre-transplant on Day 0 at a dose of 1g orally twice a day for the duration of study follow-up (2 years after the final islet transplant).
  Other Names: Cellcept
Drug: Tacrolimus — Tacrolimus may be used only as a supplement to maintenance mycophenolate mofetil (MMF) in those cases where the trough level is below the therapeutic range. Tacrolimus will be administered orally twice a day to maintain trough levels of 3-5 ng/mL. Generic equivalents of Prograf® will not be permitted.
  Other Names: Prograf
Procedure: Intraportal infusion of islet cells — The infusion of allogeneic pancreatic islet cells (islet transplant[s]) will occur intraportally.

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to determine the safety and effectiveness of islet transplantation using a steroid-free, calcineurin-inhibitor-free belatacept based immunosuppressive medication, for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes.

DETAILED DESCRIPTION:
Type 1 diabetes is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows long-term survival in individuals with type 1 diabetes; however, it does not guarantee constant normal blood sugar control. Because of this, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure. Some individuals with type 1 diabetes develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, transplantation of pancreatic islets is a possible treatment option. Unfortunately, insulin independence among islet transplant recipients tends to decline over time. New strategies aimed at promoting engraftment of transplanted islets are needed to improve the clinical outcomes associated with this procedure. The purpose of this study is determine the safety and efficacy of islet transplantation, when combined with an immunosuppressive medication regimen containing belatacept, for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes. This study will also seek to improve the understanding of determinants of success and failure of islet transplants for type 1 diabetes.

Eligible participants will be randomly assigned to this study or a site-specific Phase 3 islet transplantation study (CIT-07). Participants in this study will receive up to three separate islet transplants and a regimen of immunosuppressive medications consisting of belatacept, basiliximab (an IL-2 monoclonal antibody receptor blocker), and mycophenolate mofetil. Participants will begin receiving all three drugs on the day of the first islet transplant. Belatacept will also be administered again on Days 4, 14, 28, 56, and 84 post-transplant and then every 4 weeks for the duration of the study.

If the participant receives daclizumab, it will also be given again on Days 14, 28, 42, and 56 post-transplant; if the participant receives basiliximab, it will also be given again on Day 4 post-transplant. Mycophenolate mofetil will also be given for the duration of the study.

Transplantations will involve an inpatient hospital stay and intraportal infusion of islet cells. Participants who do not achieve or maintain insulin independence by Day 75 post-transplant will be considered for a second islet transplant. Participants who remain dependent on insulin for longer than 1 month after the second transplant and who show partial graft function will be considered for a third islet transplant. Participants who do not meet the criteria for a subsequent transplant and do not have a functioning graft will enter a reduced follow-up period.

There will be up to 25 study visits following each transplant. A physical exam, review of adverse events, and blood collection will occur at most visits. A chest x-ray, abdominal ultrasound, electrocardiogram, quality of life questionnaires, urine collection, and more extensive blood testing will occur at some visits. Participants will also test their own blood glucose levels at least five times per day throughout the study. A 24-month follow-up period will take place after the participant's last transplant.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures
* Clinical history compatible with type 1 diabetes with onset of disease at less than 40 years of age, insulin dependence for at least 5 years at study entry, and a sum of age and insulin dependent diabetes duration of at least 28
* Absent stimulated C-peptide (less than 0.3 ng/mL) 60 and 90 minutes post-mixed-meal tolerance test
* Involvement of intensive diabetes management, defined as:

  1. Self-monitoring of glucose no less than a mean of three times each day averaged over each week
  2. Three or more insulin injections each day or insulin pump therapy
  3. Under the care of an endocrinologist, diabetologist, or diabetes specialist with at least three clinical evaluations during the past 12 months prior to study enrollment
* At least one episode of severe hypoglycemia, defined as an event with one of the following symptoms: memory loss; confusion; uncontrollable behavior; irrational behavior; unusual difficulty in awakening; suspected seizure; seizure; loss of consciousness; or visual symptoms, in which the participant was unable to treat him/herself and which was associated with either a blood glucose level less than 54 mg/dL or prompt recovery after oral carbohydrate, intravenous glucose, or glucagons in the 12 months prior to study enrollment
* Reduced awareness of hypoglycemia. More information about this criterion is in the protocol.

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m^2 or weight less than or equal to 50 kg (110 lbs)
* Insulin requirement of more than 1.0 IU/kg/day or less than 15 U/day
* HbA1c greater than 10%
* Untreated proliferative diabetic retinopathy
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg
* Measured glomerular filtration rate using iohexol of less than 80 mL/min/1.73m^2.
* Presence or history of macroalbuminuria (greater than 300 mg/g creatinine)
* Presence or history of panel-reactive anti-Histocompatibility Antigen (HLA) antibody levels greater than background by flow cytometry. More information about this criterion is in the protocol.
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and 4 months after study completion
* All women more than 35 years and women of any age who have first degree relatives with a history of breast carcinoma or who have other risk factors of breast carcinoma. More information about this criterion is in the study protocol.
* Active infection, including hepatitis B, hepatitis C, human immunodeficiency virus (HIV). Presence or history of tuberculosis. More information about these criteria is in the protocol.
* Negative for Epstein-Barr virus (EBV) by anti-viral capsid antigen (VCA) IgG (EBV VCA-IgG) determination
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection in the past year
* History of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Baseline Hgb below the lower limits of normal, lymphopenia, neutropenia, or thrombocytopenia
* History of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or individuals with an international normalized ratio (INR) greater than 1.5.
* Severe coexisting cardiac disease, defined as:

  1. Heart attack within the last 6 months
  2. Evidence of ischemia on functional heart exam within the year prior to study entry
  3. Left ventricular ejection fraction less than 30%
* Persistent elevation of liver function tests at study entry
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy, defined as fasting LDL cholesterol greater than 130 mg/dL and/or fasting triglycerides greater than 200 mg/dL
* Currently receiving treatment for a medical condition that requires chronic use of systemic steroids except for the use of 5 mg or less of prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only
* Treatment with any antidiabetic medication other than insulin within the past 4 weeks
* Previous receipt of belatacept
* Use of any investigational agents within the past 4 weeks
* Received a live attenuated vaccine(s) within the past 2 months
* Any medical condition that, in the opinion of the investigator, might interfere with safe participation in the trial

  * Treatment with any immunosuppressive regimen at the time of enrollment.
  * A previous islet transplant.
  * A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and the transplant occurred more than 6 months prior to enrollment.
* Known hypersensitivity to mycophenolate mofetil or any of its components
* Imprisonment or involuntary incarceration for treatment of either a psychiatric or physical illness
* Rare hereditary deficiency of hypoxanthine-guanine phosphoribosyltransferase (HGPRT) such as Lesch-Nyhan and Kelly-Seegmiller syndrome
* Dietary restriction of phenylalanine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with insulin independence | 75 days after first islet transplant

SECONDARY OUTCOMES:
Proportion of subjects with an HbA1c <7.0% AND free of severe hypoglycemic events | from Day 28 to Day 365, inclusive, after the first islet transplant
Proportion of subjects with an HbA1c <7.0% AND free of severe hypoglycemic events | from Day 28 to Day 365, inclusive, after the final islet transplant
Percent reduction in insulin requirements, HbA1c, Mean amplitude of glycemic excursions (MAGE), Glycemic lability index (LI), Ryan hypoglycemia severity (HYPO) score | 75 Days after first and final islet transplant
Basal (fasting) and 90-min glucose and C-peptide derived from the mixed-meal tolerance test (MMTT), beta-score, C-peptide: glucose-creatinine ration, acute insulin response to glucose | 75 Days after first and final islet transplant
Insulin sensitivity and disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance test (FSIGT) test | 75 days after first and final islet transplant
Glucose variability and hypoglycemia duration, derived from the continuous glucose monitoring system (CGMS), quality of life (QOL) measures | 75 days after first and final islet transplant
Percent reduction in insulin requirements, HbA1c, Mean amplitude of glycemic excursions (MAGE), Glycemic lability index (LI), Clarke Score, Ryan hypoglycemia severity (HYPO) score | 365 days after first and final islet transplant
Basal (fasting) and 90-min glucose and C-peptide derived from the mixed-meal tolerance test (MMTT), beta-score, C-peptide: glucose-creatinine ratio | 365 days after first and final islet transplant
Insulin sensitivity and disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance test (FSIGT) test | 365 days after first and final islet transplant
Glucose variability and hypoglycemia duration, derived from the continuous glucose monitoring system (CGMS), quality of life (QOL) measures | 365 days after first and final islet transplant
Proportion of participants receiving a second or third islet transplant | 365 days after first and final islet transplant
Rate of favorable outcome at each center preparing islets (rate of subjects with an HbA1c < 7.0% and free of severe hypoglycemic events) | 365 days after first and final islet transplant
Incidence and severity of adverse events related to the islet transplant procedure | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence and severity of adverse events related to immunosuppression therapy | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence of change in the immunosuppression drug regimen | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence of immune sensitization defined by presence of Histocompatibility Antigen (HLA) antibodies absent prior to transplantation | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence of worsening retinopathy | 365 days following the first islet transplant
Percent reduction in insulin requirements, HbA1c, Mean amplitude of glycemic excursions (MAGE), Glycemic lability index (LI), Clarke Score, Ryan hypoglycemia severity (HYPO) score | From 75 days to 365 days after final islet transplant
Basal (fasting) and 90-min glucose and C-peptide derived from the mixed-meal tolerance test (MMTT), beta-score, C-peptide: glucose-creatinine ratio | From 75 days to 365 days after final islet transplant
Insulin sensitivity and disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance test (FSIGT) test | From 75 days to 365 days after final islet transplant
Glucose variability and hypoglycemia duration, derived from the continuous glucose monitoring system (CGMS), quality of life (QOL) measures | From 75 days to 365 days after final islet transplant
Proportion of participants receiving a second or third islet transplant | From 75 days to 365 days after final islet transplant
Rate of favorable outcome at each center preparing islets (rate of subjects with an HbA1c < 7.0% and free of severe hypoglycemic events) | From 75 days to 365 days after final islet transplant
Percent reduction in insulin requirements, number of severe hypoglycemic events from 28 days to 2 years, HbA1c, Clarke Score | Two years after final islet transplant
Basal (fasting) and 90-min glucose and C-peptide derived from the mixed-meal tolerance test (MMTT), beta-score, C-peptide | Two years after final islet transplant
Glucose variability and hypoglycemia duration, derived from the continuous glucose monitoring system (CGMS), quality of life (QOL) measures | Two years after final islet transplant
Safety associated with conventional immunosuppression | Two years after final islet transplant
Renal function as measured by serum creatinine, glomerular filtration rate (GFR) and other relevant laboratory parameters | Two years after final islet transplant
Lipid profiles (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol) | Two years after final islet transplant

CONTACTS AND LOCATIONS:
Overall Officials: A.M. James Shapiro, MD, PhD, Study Chair — Clinical Islet Transplant Program, University of Alberta; Nicole Turgeon, MD, Study Chair — Clinical Islet Transplant Program, Emory University
Locations (2):
- Emory University, Atlanta, Georgia, United States
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Gala-Lopez B, Kin T, O'Gorman D, Pepper AR, Senior P, Humar A, Shapiro AM. Microbial contamination of clinical islet transplant preparations is associated with very low risk of infection. Diabetes Technol Ther. 2013 Apr;15(4):323-7. doi: 10.1089/dia.2012.0297. Epub 2013 Feb 25. PMID 23438305
- See also: Click here for the Clinical Islet Transplantation Consortium Web site — http://www.citisletstudy.org
- See also: National Institute of Allergy and Infectious Diseases — http://www.niaid.nih.gov/Pages/default.aspx